CLINICAL TRIAL: NCT06824194
Title: A Phase 3, Randomized, Modified Double-blind, Active-controlled, Parallel-group, 2 Arm Study to Investigate the Safety of a 4-dose Regimen of a 21-valent Pneumococcal Conjugate Vaccine in Healthy Infants and Toddlers
Brief Title: Study of the Safety of a 21-valent Pneumococcal Conjugate Vaccine in Healthy Infants From Approximately 2 Months of Age
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PSK05; U1111-1295-5983 (Other: WHO ICTRP)
Record Dates: First submitted 2025-02-07; First posted 2025-02-13 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Pneumococcal Immunization
MeSH Terms: interventions — RIX4414 vaccine; RotaTeq; Vaxelis; Chickenpox Vaccine; Measles-Mumps-Rubella Vaccine; Hepatitis A Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Modified double-blind
  * Blinding for vaccine group assignment: participants and participant's parent(s) / legally acceptable representative(s) (LARs), outcome assessors, Investigators, laboratory personnel, and Sponsor study staff
  * No blinding for vaccine group assignment: those preparing and administering the study interventions
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1: PCV21 (Experimental): Participants will be administered via intramuscular injection (IM) a 4-dose PCV21 regimen at approximately 2, 4, 6 and 12 to 15 MoA
  Interventions: Biological: PCV21 vaccine; Biological: M-M-R II vaccine; Biological: Rotarix; Biological: RotaTeq; Biological: Vaxelis vaccine; Biological: Varivax; Biological: Priorix; Biological: VAQTA; Biological: Havrix
- Group 2: 20vPCV (Active Comparator): Participants will be administered via intramuscular injection (IM) a 4-dose 20vPCV regimen at approximately 2, 4, 6 and 12 to 15 MoA
  Interventions: Biological: Prevnar 20 vaccine; Biological: M-M-R II vaccine; Biological: Rotarix; Biological: RotaTeq; Biological: Vaxelis vaccine; Biological: Varivax; Biological: Priorix; Biological: VAQTA; Biological: Havrix

INTERVENTIONS:
Biological: PCV21 vaccine — Pharmaceutical form:Suspension for injection-Route of administration:Intramuscular
  Other Names: 515
  Arms: Group 1: PCV21
Biological: Prevnar 20 vaccine — Pharmaceutical form:Suspension for injection-Route of administration:Intramuscular
  Other Names: Prevnar20™
  Arms: Group 2: 20vPCV
Biological: M-M-R II vaccine — Pharmaceutical form:Powder, lyophilized, for suspension for reconstitution-Route of administration:Subcutaneous or Intramuscular
  Other Names: M-M-R™ II
Biological: Rotarix — Pharmaceutical form:Solution-Route of administration:Oral
  Other Names: Rotarix™
Biological: RotaTeq — Pharmaceutical form:Solution-Route of administration:Oral
  Other Names: RotaTeq™
Biological: Vaxelis vaccine — Pharmaceutical form:Suspension for injection-Route of administration:Intramuscular
  Other Names: Vaxelis™
Biological: Varivax — Pharmaceutical form:Powder, lyophilized, for suspension for reconstitution-Route of administration:Subcutaneous or Intramuscular
  Other Names: Varivax™
Biological: Priorix — Pharmaceutical form:Lyophilized, for suspension for reconstitution-Route of administration:Subcutaneous
  Other Names: Priorix™
Biological: VAQTA — Pharmaceutical form:Suspension for Injection-Route of administration:Intramuscular
  Other Names: VAQTA™
Biological: Havrix — Pharmaceutical form:Suspension for Injection-Route of administration:Intramuscular
  Other Names: Havrix™

SUMMARY:
This study is a Phase 3, randomized, modified double-blind study which aims to document the safety profile of the PCV21 vaccine (investigational pneumococcal vaccine) compared to a licensed 20-valent pneumococcal conjugate vaccine in infants aged from approximately 2 months (42 to 89 days).

The study duration per participant will be up to approximately 19 months. The study vaccines (either PCV21 or 20vPCV) will be administered at approximately 2, 4, 6 and 12 to 15 months of age. Routine pediatric vaccines will be given as per local recommendations.

There will be 6 study visits:

Visit (V)01, V02 separated from V01 by 60 days, V03 separated from V02 by 60 days, V04 separated from V03 by 30 days, V05 at 12 months of age until 15 months of age, V06 separated from V05 by 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Aged 42 to 89 days on the day of inclusion
* Participants who are healthy as determined by medical evaluation including medical history and physical examination
* Born at full term of pregnancy (≥ 37 weeks) and with a birth weight ≥ 2.5 kg or born after a gestation period above 28 (> 28 weeks) through 36 weeks with a birth weight ≥ 1.5 kg, and in both cases medically stable as assessed by the investigator

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy; or long-term systemic corticosteroid therapy
* History of microbiologically confirmed Streptococcus pneumoniae infection or disease
* Any contraindication to the routine pediatric vaccine being administered in the study
* History of seizure or significant stable or progressive neurologic disorders such as infantile spasms, inflammatory nervous system diseases, encephalopathy, cerebral palsy
* Known systemic hypersensitivity to any of the study interventions components, or history of a life-threatening reaction to the study interventions used in the study or to a product containing any of the same substances
* Laboratory-confirmed or known thrombocytopenia, as reported by the parent(s) / legal acceptable representative (LAR(s)), contraindicating intramuscular (IM) injection
* Bleeding disorder, or receipt of anticoagulants in the 3 weeks preceding inclusion, contraindicating IM injection
* Chronic illness that, in the opinion of the investigator, is at a stage where it might interfere with study conduct or completion
* Moderate or severe acute illness/infection (according to investigator judgment) or febrile illness (temperature ≥ 38.0°C [≥ 100.4°F]) on the day of study intervention administration. A prospective participant should not be included in the study until the condition has resolved or the febrile event has subsided
* Receipt of any non-US Food and Drug Administration (FDA) approved vaccine in the 4 weeks preceding the study intervention administration or planned receipt of any non-US FDA approved vaccine in the 4 weeks following the study intervention administration, including monovalent pandemic influenza vaccines and multivalent influenza vaccines, as applicable per local recommendations.
* Receipt of any Bacillus of Calmette and Guerin (BCG) vaccine within 4 weeks preceding the first study intervention administration or planned receipt any BCG vaccine within the study period
* Previous vaccination against S. pneumoniae
* Previous vaccination against the following antigens: diphtheria, tetanus, pertussis, H. influenzae type b, poliovirus
* Receipt of more than 1 dose of hepatitis B vaccine
* Receipt of immune globulins, blood or blood-derived products since birth
* Participation at the time of study enrollment (or in the 6 weeks preceding the first study intervention administration) or planned participation during the present study period in another clinical study investigating a vaccine, drug, medical device, or medical procedure

Note: The above information is not intended to contain all considerations relevant to a potential participation in a clinical trial.

Ages: 42 Days to 89 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2320 (Estimated)
Dates: Start 2025-02-18 (Actual); Primary Completion 2027-05-12 (Estimated); Study Completion 2027-05-12 (Estimated)

PRIMARY OUTCOMES:
Presence of any immediate adverse events (AEs) | Within 30 minutes after each vaccination
  Number of participants experiencing solicited and unsolicited immediate AEs
Presence of solicited injection site and systemic reactions through 7 days after each vaccine injection | Through 7 days after each vaccine injection
  Number of participants experiencing solicited injection site and systemic reactions
Presence of unsolicited (spontaneously reported) injection site reactions and unsolicited systemic AEs through 30 days after each vaccine injection | Through 30 days after each vaccine injection
  Number of participants experiencing unsolicited injection site reactions and unsolicited systemic AEs
Presence of serious adverse events (SAEs) throughout the study (through 6 months post- last vaccine injection) | Throughout the study (through 6 months post-last vaccine injection), approximately 19 months
  Number of participants experiencing SAEs
Presence adverse events of special interest (AESIs) throughout the study (through 6 months post- last vaccine injection) | Throughout the study (through 6 months post-last vaccine injection), approximately 19 months
  Number of participants experiencing AESIs

CONTACTS AND LOCATIONS:
Locations (124):
- United States (97):
  - Alabama Clinical Therapeutics - Birmingham - St. Vincent's Drive- Site Number : 8400013, Birmingham, Alabama
  - University of Alabama at Birmingham- Site Number : 8400130, Birmingham, Alabama
  - Lakeview Clinical Research- Site Number : 8400054, Guntersville, Alabama
  - Midway Medical Clinic- Site Number : 8400091, Oneonta, Alabama
  - Noble Clinical Research- Site Number : 8400121, Tucson, Arizona
  - The Children's Clinic- Site Number : 8400079, Jonesboro, Arkansas
  - Helios CR, Inc. - Little Rock- Site Number : 8400090, Sherwood, Arkansas
  - Helping Hands Healthcare Group - Fullerton- Site Number : 8400063, Fullerton, California
  - Advanced Investigative Medicine- Site Number : 8400055, Hawthorne, California
  - Matrix Clinical Research - Los Angeles- Site Number : 8400026, Los Angeles, California
  - Alliance Research Institute - Lynwood- Site Number : 8400099, Lynwood, California
  - Madera Family Medical Group- Site Number : 8400011, Madera, California
  - FOMAT-Golden Valley Health Centers- Site Number : 8400084, Merced, California
  - Stanford University Medical Center CTRU - 800 Welch Road- Site Number : 8400072, Palo Alto, California
  - Center for Clinical Trials - Paramount- Site Number : 8400100, Paramount, California
  - Integrated Clinical Research LLC- Site Number : 8400027, Sherman Oaks, California
  - Emanate Health - Queen of the Valley Hospital- Site Number : 8400105, West Covina, California
  - All in One Clinic- Site Number : 8400127, Whittier, California
  - Amicis Research Center-Winnetka- Site Number : 8400128, Winnetka, California
  - Emerson Clinical Research Institute - Washington - Connecticut Avenue- Site Number : 8400102, Washington D.C., District of Columbia
  - D&H Doral Research Center- Site Number : 8400095, Doral, Florida
  - Nextlevel Research Center- Site Number : 8400065, Doral, Florida
  - PAS RESEARCH-Lutz- Site Number : 8400103, Lutz, Florida
  - Abba Medical Research- Site Number : 8400064, Miami, Florida
  - D&H National Research Center- Site Number : 8400085, North Miami, Florida
  - Alfa Medical Research LLC- Site Number : 8400111, Pembroke Pines, Florida
  - PAS Research - Tampa- Site Number : 8400113, Tampa, Florida
  - Morehouse School of Medicine - Atlanta- Site Number : 8400093, Atlanta, Georgia
  - Primary Pediatrics of Macon at Velocity Clinical Research- Site Number : 8400004, Macon, Georgia
  - CenExel - iResearch - Savannah- Site Number : 8400057, Savannah, Georgia
  - Bingham Memorial Hospital - Blackfoot- Site Number : 8400114, Blackfoot, Idaho
  - Elite Clinical Trials - Blackfoot- Site Number : 8400017, Blackfoot, Idaho
  - Clinical Research Prime- Site Number : 8400022, Idaho Falls, Idaho
  - Eagle Clinical Research- Site Number : 8400087, Chicago, Illinois
  - University of Chicago Medical Center- Site Number : 8400062, Chicago, Illinois
  - MidValley Research - Moline- Site Number : 8400096, Moline, Illinois
  - South Bend Clinic - Main Campus- Site Number : 8400023, South Bend, Indiana
  - Integrated Clinical Trial Services- Site Number : 8400059, West Des Moines, Iowa
  - Kentucky Pediatric Research- Site Number : 8400014, Bardstown, Kentucky
  - University of Kentucky Chandler Medical Center- Site Number : 8400034, Lexington, Kentucky
  - Novak Center For Children's Health- Site Number : 8400073, Louisville, Kentucky
  - Bluegrass Clinical Research - Louisville - Blankenbaker Parkway- Site Number : 8400056, Louisville, Kentucky
  - Velocity Clinical Research - Lafayette- Site Number : 8400046, Lafayette, Louisiana
  - Research Works INC- Site Number : 8400035, New Orleans, Louisiana
  - The Pediatric Center- Site Number : 8400075, Columbia, Maryland
  - The Pediatric Center of Frederick- Site Number : 8400074, Frederick, Maryland
  - Virgo Carter Pediatrics- Site Number : 8400001, Silver Spring, Maryland
  - Michigan Institute of Research- Site Number : 8400131, Allen Park, Michigan
  - Vida Clinical Studies - Dearborn- Site Number : 8400094, Dearborn, Michigan
  - Clinical Research Institute - Minneapolis- Site Number : 8400002, Minneapolis, Minnesota
  - Jefferson City Medical Group- Site Number : 8400129, Jefferson City, Missouri
  - Midwest Children's Health Research Institute - Lincoln - Salt Creek Circle- Site Number : 8400019, Lincoln, Nebraska
  - Midwest Children's Health Research Institute- Site Number : 8400016, Lincoln, Nebraska
  - Be Well Clinical Studies - Lincoln- Site Number : 8400031, Lincoln, Nebraska
  - Midwest Childrens Health Research Institute- Site Number : 8400021, Lincoln, Nebraska
  - Midwest Children's Health Research Institute - Lincoln - West A Street- Site Number : 8400045, Lincoln, Nebraska
  - PAS Research - Henderson- Site Number : 8400033, Henderson, Nevada
  - SUNY Downstate Medical Center- Site Number : 8400039, Brooklyn, New York
  - Child Health Care Associates - East Syracuse- Site Number : 8400005, East Syracuse, New York
  - GRO Clinical- Site Number : 8400109, Hyde Park, New York
  - PAS Research-Bronx- Site Number : 8400104, The Bronx, New York
  - Advantage Clinical Trials- Site Number : 8400030, The Bronx, New York
  - Atrium Health - Myers Park- Site Number : 8400080, Charlotte, North Carolina
  - Atrium Health - STRIVE Vaccine Research Clinic- Site Number : 8400060, Charlotte, North Carolina
  - Haywood Pediatric and Adolescent Medicine Group- Site Number : 8400051, Clyde, North Carolina
  - East Carolina University- Site Number : 8400061, Greenville, North Carolina
  - Piedmont Healthcare - Family Medicine- Site Number : 8400077, Statesville, North Carolina
  - Legacy Clinical Trials Oklahoma City- Site Number : 8400097, Oklahoma City, Oklahoma
  - Cyn3rgy Research- Site Number : 8400029, Gresham, Oregon
  - Kid's Way Pediatrics- Site Number : 8400119, Hermitage, Pennsylvania
  - Pas Research - Pittsburgh- Site Number : 8400050, Pittsburgh, Pennsylvania
  - Neighbors Pediatrics- Site Number : 8400068, Charleston, South Carolina
  - Tribe Clinical Research - Simpsonville- Site Number : 8400069, Simpsonville, South Carolina
  - Parkside Pediatrics - Simpsonville- Site Number : 8400078, Simpsonville, South Carolina
  - Tribe Clinical Research - Spartanburg- Site Number : 8400083, Spartanburg, South Carolina
  - Austin Regional Clinic - ARC Four Points- Site Number : 8400082, Austin, Texas
  - Cedar Health Research - Dallas- Site Number : 8400092, Dallas, Texas
  - PAS Research - Children's Care Clinic- Site Number : 8400012, Edinburg, Texas
  - The University of Texas Health Science Center- Site Number : 8400024, Houston, Texas
  - Mercury Clinical Research - Houston - Savoy Drive- Site Number : 8400049, Houston, Texas
  - Pediatric Associates - Houston- Site Number : 8400101, Houston, Texas
  - GLRI - McAllen Research- Site Number : 8400098, Pharr, Texas
  - AIM Trials- Site Number : 8400052, Plano, Texas
  - Helios Clinical Research - Plano- Site Number : 8400009, Plano, Texas
  - Tekton Research - FM78- Site Number : 8400003, San Antonio, Texas
  - North Houston Internal Medicine & Pediatric Clinic- Site Number : 8400018, Tomball, Texas
  - Wee Care Pediatrics - Kaysville- Site Number : 8400028, Kaysville, Utah
  - Wee Care Pediatrics - Layton- Site Number : 8400044, Layton, Utah
  - Rio Clinical Trials - Canyon View- Site Number : 8400132, Ogden, Utah
  - Utah Valley Pediatrics - Orem- Site Number : 8400053, Orem, Utah
  - Ogden Clinic - Mountain View - CCT Research- Site Number : 8400032, Pleasant View, Utah
  - Pediatric Care - Provo- Site Number : 8400041, Provo, Utah
  - Wee Care Pediatrics - Roy- Site Number : 8400070, Roy, Utah
  - J. Lewis Research - Foothill Family Clinic - Salt Lake City- Site Number : 8400058, Salt Lake City, Utah
  - Wee Care Pediatrics - Syracuse- Site Number : 8400066, Syracuse, Utah
  - National Clinical Research- Site Number : 8400010, Richmond, Virginia
  - Full Circle Family Medicine- Site Number : 8400110, Germantown, Wisconsin
- Honduras (3):
  - Investigational Site Number : 3400001, San Pedro Sula
  - Investigational Site Number : 3400002, Tegucigalpa
  - Investigational Site Number : 3400003, Tegucigalpa
- Mexico (6):
  - Investigational Site Number : 4840003, León, Guanajuato
  - Investigational Site Number : 4840001, Mexico City, Mexico City
  - Investigational Site Number : 4840007, Morelia, Michoacán
  - Investigational Site Number : 4840009, Cuernavaca, Morelos
  - Investigational Site Number : 4840002, Temixco, Morelos
  - Investigational Site Number : 4840008, Ecatepec de Morelos
- Puerto Rico (6):
  - Investigational Site Number : 6300001, Bayamón
  - Investigational Site Number : 6300002, Bayamón
  - Investigational Site Number : 6300005, Guayama
  - Investigational Site Number : 6300004, Ponce
  - Investigational Site Number : 6300003, San Juan
  - Investigational Site Number : 6300006, San Juan
- Thailand (3):
  - Investigational Site Number : 7640002, Bangkok
  - Investigational Site Number : 7640001, Chiang Mai
  - Investigational Site Number : 7640003, Hat Yai
- Turkey (Türkiye) (9):
  - Investigational Site Number : 7920004, Ankara
  - Investigational Site Number : 7920002, Ankara
  - Investigational Site Number : 7920006, Ankara
  - Investigational Site Number : 7920003, Istanbul
  - Investigational Site Number : 7920007, Istanbul
  - Investigational Site Number : 7920009, Izmir
  - Investigational Site Number : 7920005, Izmir
  - Investigational Site Number : 7920008, Izmir
  - Investigational Site Number : 7920010, Trabzon

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: PSK05 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=26405&tenant=MT_SNY_9011